CLINICAL TRIAL: NCT02739360
Title: An Open Label, Roll Over Study to Provide Idelalisib to Subjects Previously Treated With the Investigational PI3Kδ Inhibitor, GS-9820
Brief Title: Roll Over Study to Provide Idelalisib to Participants Previously Treated With the Investigational PI3Kδ Inhibitor, GS-9820
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-313-2120; 2015-005766-39 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-01

CONDITIONS: Lymphoid Malignancies
MeSH Terms: interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Idelalisib (Experimental): Participants will receive idelalisib until unacceptable toxicity, disease progression, study discontinuation, or death occurs.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg tablet administered orally twice daily
  Other Names: Zydelig®

SUMMARY:
The primary objective of this study is to provide idelalisib to participants receiving GS-9820 in Gilead-sponsored Study GS-US-315-0102 at the time of study closure.

ELIGIBILITY:
Key Inclusion Criteria:

* Receiving GS-9820 in Study GS-US-315-0102 with objective evidence of clinical benefit
* Evidence of a personally signed informed consent

Key Exclusion Criteria:

* Known hypersensitivity or intolerance to any of the active substances or excipients in the formulation of idelalisib
* Toxicities that would preclude initiating therapy with idelalisib prior to enrollment
* Concurrent participation in another therapeutic clinical trial
* Ongoing infection, treatment, or prophylaxis for cytomegalovirus (CMV) within the past 28 days.

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the Netherlands. The first participant was screened on 04 May 2016. The last study visit occurred on 28 December 2017.
Pre-assignment Details: Six participants previously enrolled in Study GS-US-315-0102 were offered screening for enrollment into this study.
Period: Overall Study
Arm/Group | Idelalisib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Study terminated by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug.
Arm/Group | Idelalisib
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  From 65 - 84 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-Emergent ≥ Grade 3 Adverse Events, Serious Adverse Events (SAEs), and Deaths
Description: The severity of Adverse Events were graded using the Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03. An SAE was defined as an event that, at any dose, resulted in one or more of the following: 1) Death, 2) Life-threatening, 3) In-patient hospitalization or prolongation of existing hospitalization, 4) Persistent or significant disability/incapacity, 5) A congenital anomaly/birth defect, or 6) A medically important event or reaction.
Time Frame: Up to Day 602 plus 30 days
Population: Safety Analysis Set: participants who took at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 3
Participants
  ≥ Grade 3 Adverse Event | 1
  SAE | 1
  Death | 0

ADVERSE EVENTS:
Time Frame: Up to Day 602 plus 30 days
Description: Safety Analysis Set: participants who took at least 1 dose of study drug.
Arm/Group | Idelalisib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=3)
Cholangitis (Hepatobiliary disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=3)
Anaemia (Blood and lymphatic system disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Aspartate aminotransferase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Intermittent claudication (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02739360/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT02739360/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02739360/Prot_002.pdf
  • Study Protocol: Amendment 3 (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT02739360/Prot_003.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT02739360/SAP_004.pdf